CLINICAL TRIAL: NCT05126797
Title: 3D Printed Oral Stents for Patients Receiving Head and Neck Radiation Therapy
Brief Title: 3D Printed Oral Stents for Patients With Head and Neck Cancer Receiving Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrativley Complete, <75% Participants
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2017-0269; NCI-2019-02460 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0269 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-03; First posted 2021-11-19 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Malignant Head and Neck Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 3D printed stent+ MDASI-3D Oral Stents Questionnaire (Other): Patients wear a customized 3D printed oral stent over 5-10 minutes in the supine position at the time of radiation simulation, before starting radiation therapy, and in the 3rd to 5th week of radiation therapy. Patients may also optionally wear the commercially-made stent called TruGuard at these timepoints. Ancillary Studies (MDASI-3D Oral Stents Questionnaire)
  Interventions: Other: Questionnaire Administration; Device: Stent Device

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Device: Stent Device — Wear customized 3D printed oral stent
  Other Names: Stent

SUMMARY:
This trial studies how a customized 3D-printed oral stent compares to a standard stent made by a dentist for use in imaging scans in patients with head and neck cancer receiving radiation therapy. Oral stents are designed to help prevent radiation-related side effects while receiving radiation therapy. Traditional oral stents are created by dentists, require at least 2 separate appointments, and may not be as cost-effective. A customized, 3D-printed oral stent may perform as well as a standard stent made by a dentist and have a significantly shorter turnaround to device delivery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether a customized 3 dimensional (3D) printed oral stent achieves non-inferior levels of patient reported outcomes as the standard dental-fabricated oral stents at the time prior to starting treatment.

SECONDARY OBJECTIVES:

I. To evaluate the performance of the 3D stent on imaging parameters (i.e. mandibular and soft tissue displacement) for degree of normal tissue sparing.

II. Evaluate the levels of patient reported outcomes after patients have developed side effects from radiation treatment.

III. To evaluate the commercially available TruGuard oral cavity positioning system.

OUTLINE:

Patients wear a customized 3D printed oral stent over 5-10 minutes in the supine position at the time of radiation simulation, before starting radiation therapy, and in the 3rd to 5th week of radiation therapy. Patients may also optionally wear the commercially-made stent called TruGuard at these timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Patient is dispositioned to receive definitive or adjuvant radiotherapy for treatment of a diagnosed head and neck malignancy.
* Treating radiation oncologist has determined the necessity of an oral stent and a device has been fabricated by dentistry at MD Anderson Cancer Center (MDACC).
* Patient has received pre-treatment imaging which includes the mandibular and maxillary dentition.
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0-2.
* Signed study-specific consent form.

Exclusion Criteria:

* No pre-treatment computed tomography (CT) imaging including the maxilla and mandible is available.
* Prior head and neck radiotherapy.
* Severe trismus with an incisal opening of < 10 mm.
* Inability to comply with the study procedures.
* Patients who have received dental stents fabricated outside of MDACC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
To evaluate whether a customized 3 dimensional (3D) printed oral stent achieves non-inferior levels of patient reported outcomes as the standard dental-fabricated oral stents at the time prior to starting treatment. | up to 2 months
  The patient will fill out a questionnaire that measures the form and fit of the 3D printed oral stent at specified time points, and this measurement will be compared with a standard stent. Score ranges(0-10) 0 None at all-10 As bad as you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Koay, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org